CLINICAL TRIAL: NCT01821391
Title: Multi-centre, Randomized, Investigator-blind, Intra-individual Active and Vehicle-controlled Study, Comparing Metvix Natural Daylight Photodynamic Therapy Versus Metvix Conventional Photodynamic Therapy in Subjects With Actinic Keratosis
Brief Title: Phase 3b Study of Metvix NDL-PDT Versus Metvix c-PDT in Subjects With Actinic Keratoses
Acronym: COMET2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.29112
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2018-02

CONDITIONS: Actinic Keratoses
Keywords: actinic keratoses; photodynamic therapy; natural daylight
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: 2 intra-individual groups:
  * Metvix NDL-PDT / Metvix c-PDT
  * Metvix NDL-PDT / Placebo c-PDT
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NDL-PDT/c-PDT (Experimental): Metvix natural daylight photodynamic therapy and Metvix conventional photodynamic therapy
  Interventions: Drug: NDL-PDT; Drug: c-PDT
- NDL-PDT/placebo c-PDT (Experimental): Metvix natural daylight photodynamic therapy and Metvix-placebo conventional photodynamic therapy
  Interventions: Drug: NDL-PDT; Drug: placebo c-PDT

INTERVENTIONS:
Drug: NDL-PDT — Metvix natural daylight photodynamic therapy
  Other Names: Metvix NDL-PDT
Drug: c-PDT — Metvix conventional photodynamic therapy
  Other Names: Metvix c-PDT
  Arms: NDL-PDT/c-PDT
Drug: placebo c-PDT — Metvix placebo conventional photodynamic therapy
  Other Names: Metvix placebo c-PDT
  Arms: NDL-PDT/placebo c-PDT

SUMMARY:
This study was to be conducted as a multi-centre, randomized, investigator-blinded, active and vehicle-controlled, intra-individual (split-face/scalp) non-inferiority (regarding efficacy) and superiority (regarding pain) study.

The primary purpose of this study is to demonstrate the non-inferiority of NDL-PDT compared to c-PDT in terms of lesion complete response rate.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild (Grade 1) and/or moderate (Grade 2) AKs on the face or the scalp on treated areas
* Subject with two symmetrical treated areas half scalps or two half faces excluding ears, chin, bridge of the nose, eyelids and lips inside the vermillion border): no more than a twofold difference in terms of total number of lesions between the two TAs

Exclusion Criteria:

* Subject with clinical diagnosis of at least one severe (Grade 3) AK on treated areas
* Subject with pigmented AK on the treated areas
* Immuno-compromised Subject for idiopathic, disease specific or therapeutic reasons
* Subject with porphyria,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Basset Seguin, PhD, MD, Principal Investigator — Hopital Saint Louis France; Bibiana Perez Garcia, MD, Principal Investigator — Hospital Ramón y Cajal Spain; Rianne Gerritsen, PhD, MD, Principal Investigator — Radboud University, Nijmegen Medical Center The Netherlands; Rolf-Markus Sziemies, PhD, MD, Principal Investigator — Klinik fur Dermatologie und Allergologie Germany; Ingrid Synnerstad, PhD, MD, Principal Investigator — Hudmottagningen Sweden
Locations (18):
- France (5):
  - Investigative site, Montpellier
  - Investigational site, Nantes
  - Investigational site, Nice
  - Investigational site, Paris
  - Investigative site, Rennes
- Germany (4):
  - Investigational site, Aachen
  - Investigational site, Berlin
  - Investigational site, Münster
  - Investigational site, Recklinghausen
- Netherlands (3):
  - Investigational site, Assen
  - Investigational site, Maastricht
  - Investigational site, Nijmegen
- Spain (4):
  - Investigational site, Huesca
  - Investigational site, Madrid
  - Investigative site, Pamplona
  - Investigational site, Valencia
- Sweden (2):
  - Investigational site, Karlskoga
  - Investigational site, Norrköping

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Participants applied single dose of Metvix cream topically followed by NDL-PDT (test treatment) on one half-face/scalp and on the contra-lateral side of face/scalp applied Metvix cream topically followed by c- PDT (active comparator) on Day 0 (Baseline).
- Group 2: Participants applied a single dose of Metvix cream topically followed by NDL-PDT (test treatment) on one half-face/scalp and on the contra-lateral side of face/scalp applied Metvix vehicle cream (placebo) followed by c-PDT on Day 0 (Baseline).
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 108 | 23
Completed | 107 | 23
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 108 | 23 | 131
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0 | 0 | 0
  Age: Between 18 and 65 years | 19 | 2 | 21
  Age: >=65 years | 89 | 21 | 110
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 10
  Male | 99 | 22 | 121
Race [Count of Participants; unit: Participants]
  White | 108 | 22 | 130
  Other | 0 | 1 | 1
Phototype [Count of Participants; unit: Participants] — Fitzpatrick skin phototype is a system used to describe a person's skin type. It ranges from skin phototype I to III. Where, skin phototype I = pale white skin, always burns easily, never tans; skin phototype II = fair skin, always burns easily, tans minimally and with difficulty; skin phototype III = darker white skin, burns minimally, tans gradually and uniformly.
  Participants
    Phototype I | 10 | 1 | 11
    Phototype II | 69 | 17 | 86
    Phototype III | 24 | 3 | 27
    Phototype IV | 5 | 2 | 7
Duration of AK (years) [Mean (Standard Deviation); unit: years] | 9.66 (8.07) | 6.79 (5.81) | 9.15 (7.78)

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) Change From Baseline in Total Lesion Complete Response at Week 12 in Group 1
Description: The lesion complete response rate was defined as the percentage of pre-existing and treated lesions at Baseline that were assessed as clear (complete disappearance of the lesion, visually and by palpation) at Week 12. New lesions or the lesions in non-complete response were not not considered in the lesion response assessment. This outcome measure was analyzed as an intra-individual comparison between Metvix NDL-PDT on one side of the face/scalp and Metvix vehicle cream (placebo) c-PDT on the contralateral side (Group I).
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) population included entire population enrolled and randomized. ITT analysis imputed missing data using a worst case approach and considered the lesions with missed lesion response assessment as not responded (ITT/Worst-case) lesions.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- Group I: Metvix NDL-PDT: Participants applied topically a single dose of Metvix cream followed by NDL-PDT on Day 0 (Baseline).
- Group I: Metvix c-PDT: Participants applied topically a single dose of Metvix cream followed by C-PDT on Day 0 (Baseline).
Arm/Group | Group I: Metvix NDL-PDT | Group I: Metvix c-PDT
Number analyzed (Participants) | 108 | 108
percentage change from baseline | 68.4 (27.7) | 71.5 (27.6)
Statistical Analysis 1: Comparison: Group I: Metvix NDL-PDT vs Group I: Metvix c-PDT; Test type: Superiority; p = 0.2665, Paired Student's t test

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- NDL-PDT: Metvix natural daylight photodynamic therapy treated side
- c-PDT: Metvix conventional photodynamic therapy treated side
- Placebo c-PDT: Placebo conventional photodynamic therapy treated side
- Unspecific Treated Side: AE occuring outside the treated area + systemic AE
Arm/Group | NDL-PDT | c-PDT | Placebo c-PDT | Unspecific Treated Side
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/108 | 0/23 | 1/131
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/108 | 0/23 | 6/131
Other Adverse Events (participants affected / at risk) | 65/131 | 66/108 | 7/23 | 3/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NDL-PDT (N=131) | c-PDT (N=108) | Placebo c-PDT (N=23) | Unspecific Treated Side (N=131)
PULMONARY OEDEMA/ SUPPOSED WATER IN LUNG (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mallory weiss lesion in oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NDL-PDT (N=131) | c-PDT (N=108) | Placebo c-PDT (N=23) | Unspecific Treated Side (N=131)
Rash pustular (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Post procedural haemorrage (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 31 (31) | 39 (39) | 4 (4) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 8 (8) | 11 (11) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 10 (10) | 8 (8) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (13) | 16 (16) | 1 (1) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 12 (12) | 16 (17) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 12 (12) | 16 (17) | 0 (0) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No